CLINICAL TRIAL: NCT01317602
Title: Current Clinical Practice in the Management of Atrial Fibrillation in Greece: the MANAGE-AF Study
Acronym: MANAGE-AF
Status: Completed | Type: Observational
Sponsor: Hellenic Cardiovascular Research Society (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: HellenicCardiovascularRS
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multicenter, 1-year prospective, observational study of Atrial Fibrillation (AF) in Greece, designed to provide real world data regarding the characteristics of AF patients in Greece, as well as current clinical practices and adherence to the 2010 ESC guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years with any type of AF(first diagnosed, paroxysmal, persistent, long-standing persistent and permanent) according to the classification described in the recent ESC guidelines.
2. All patients should give written informed consent to participate in the study.

Exclusion Criteria:

1. Patients anticipated life expectancy less than 1 year due to a severe concomitant disease.
2. Participation in an another clinical trial, with the exception of epidemiology trials (observational) that do not influence AF management.
3. Patients with mental disability unable to comply with follow - up visits and these who are unable to provide, in written, their informed consent or patients with anticipated inability to adhere to scheduled follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The MANAGE-AF study will enroll 600 consecutive patients from the emergency cardiology departments and outpatient clinics in about 35 Greek hospitals. Their selection will be made in an effort to recruit a representative sample of patients from different geographic areas and stratums of the country.
Sampling Method: Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the management of patients with Atrial Fibrillation. | 1 year
  Evaluation of the use of anticoagulants and antithrombotic drugs. Evaluation of the doctors' compliance with the guidelines.

SECONDARY OUTCOMES:
Evaluation of the risk of strokes. | Baseline-6month-12months
  Evaluation of the risk in a large number of patients using the CHA2DS2-VASc and HAS-BLED scores.
Assessment of morbidity and mortality of patients with AF. | 1 year
  Assessment of morbidity and mortality of patients with AFduring one year follow-up in comparison with previous results from other registries.
Assessment of the compliance of patients to treatment. | Baseline-6months-12months
  Evaluation of the compliance of patients to treatment and the frequency of visits to their physician especially in terms of achieving therapeutic target INR (TTR, Time in Therapeutic Range).
Assessment of the awareness of patients about the Atrial Fibrillation. | Baseline
  Assessment of the awareness of patients about the Atrial Fibrilation and the potential risk of AF.
Assessment of patients' quality of life. | Baseline-6months-12months
  Assessment of patients' quality of life (QoL) using a specific questionnaire (EQ - 5D, http://www.euroqol.org) and EHRA score for evaluation of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Panos E. Vardas, MD, FESC, FACC, Principal Investigator — President, Hellenic Cardiovascular Research Society
Locations (27):
- Greece (27):
  - University Hospital of Alexandroupoli, Alexandroupoli
  - 7th IKA Hospital of Athens, Athens
  - Alexandra Hospital, Athens
  - Euroclinic Athens, Athens
  - General Hospital of Athens Evangelismos, Athens
  - Henry Dunant Hospital, Athens
  - KAT General Hospital, Athens
  - Korgialenio Benakio EES Hospital, Athens
  - Laiko General Hospital, Athens
  - Sismanoglio General Hospital, Athens
  - Ygeia Hospital, Athens
  - General Hospital of Chalkida, Chalcis
  - General Hospital of Chania, Chania
  - General Hospital of Chios, Chios
  - General Hospital of Edessa, Edessa
  - Thriassio General Hospital of Elefsina, Elefsina
  - University Hospital of Heraklion, Heraklion
  - General Hospital Of Heraklio Venizeleio, Heraklio
  - General Hospital of Kavala, Kavala
  - General Hospital of Komotini Sismanoglio, Komotini
  - General Hospital of Ptolemaida Mpodosakeio, Ptolemaida
  - General Hospital of Serres, Serres
  - 2nd IKA Hospital of Thessaloniki, Thessaloniki
  - Agios Loukas Clinic, Thessaloniki
  - Ippokrateio Hospital of Thessaloniki, Thessaloniki
  - University Hospital of Thessaloniki AXEPA, Thessaloniki
  - General Hospital of Volos, Volos